CLINICAL TRIAL: NCT00002039
Title: An Open Study of Foscarnet Treatment First Episode CMV-Retinitis in AIDS Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Astra USA (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 020A; 88-FOS-01
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1991-03

CONDITIONS: Cytomegalovirus Retinitis; HIV Infections
Keywords: Retinitis; AIDS-Related Opportunistic Infections; Drug Therapy, Combination; Foscarnet; Cytomegalovirus Infections; Acquired Immunodeficiency Syndrome; Antiviral Agents; Zidovudine
MeSH Terms: conditions — Cytomegalovirus Retinitis; HIV Infections; Retinitis; AIDS-Related Opportunistic Infections; Cytomegalovirus Infections; Acquired Immunodeficiency Syndrome | interventions — Foscarnet

INTERVENTIONS:
Drug: Foscarnet sodium

SUMMARY:
To evaluate the safety and efficacy of foscarnet induction therapy for treatment of AIDS patients experiencing their first episode of cytomegalovirus (CMV) retinitis. To evaluate the safety and efficacy of three different foscarnet maintenance therapy regimens. To determine the pharmacokinetics of intermittent administration of foscarnet with or without concomitant administration of zidovudine (AZT).

ELIGIBILITY:
Exclusion Criteria

Co-existing Condition:

Patients with the following are excluded:

* Any clinically significant pulmonary or neurologic impairment (e.g., patients who are intubated or comatose).
* Corneal, lens, or vitreous opacification which precludes examination of the fundi, or evidence of tuberculotic, diabetic and/or hypertensive retinopathy.
* Known allergy to foscarnet.
* Recurrent episode of cytomegalovirus (CMV) retinitis.

Concurrent Medication:

Excluded:

* Nephrotoxic drugs.

Patients with the following are excluded:

* Recurrent episode of cytomegalovirus (CMV) retinitis.
* Any clinically significant pulmonary or neurologic impairment (e.g., patients who are intubated or comatose).
* Corneal, lens, or vitreous opacification which precludes examination of the fundi, or evidence of tuberculotic, diabetic, and/or hypertensive retinopathy.
* Known allergy to foscarnet.

Prior Medication:

Excluded:

* Ganciclovir for cytomegalovirus (CMV) retinitis.
* Foscarnet for CMV retinitis.

Patients with AIDS as defined by the CDC with manifest first episode cytomegalovirus (CMV) retinitis, as identified by its characteristic ophthalmoscopic appearance and verified by fundus photography.

* Patients must be able to give informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Foscarnet Research Program / Park Plaza Hosp, Houston, Texas, United States

REFERENCES:
- [Background] Ussery FM, Karol C, Conklin R, Gathe J, Stool E, Redding K. Preliminary results from an on-going prospective evaluation of foscarnet in the treatment of AIDS-associated cytomegalovirus retinitis. Int Conf AIDS. 1989 Jun 4-9;5:551 (abstract no MCP60)